CLINICAL TRIAL: NCT01899495
Title: D1 and AT1 Receptor Interaction in Human Hypertension: Sodium Sensitivity of Blood Pressure
Brief Title: Blood Pressure Response to Sodium in the Diet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Robert M. Carey, MD, Professor of Medicine; Dean, Emeritus; University Professor Division of Endocrinology and Metabolism, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11494; P01HL074940 (NIH)
Record Dates: First submitted 2013-01-22; First posted 2013-07-15 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Hypertension
Keywords: blood pressure; hypertension; salt sensitivity
MeSH Terms: conditions — Hypertension | interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- High sodium diet and low sodium diet (Experimental): Each subject experiences both a high sodium and a low sodium diet.
  Interventions: Other: High sodium diet and low sodium diet

INTERVENTIONS:
Other: High sodium diet and low sodium diet — Isocaloric diet with 60 mEq of potassium and 1gm protein/kg body weight with high sodium 300mEq; low sodium 10 mEq.

SUMMARY:
Previous studies have demonstrated that single nucleotide polymorphisms (SNPs) of the sodium-bicarbonate co-transporter gene (SLC4A5) are associated with hypertension. We tested the hypothesis that SNPs in SLC4A5 are associated with salt sensitivity of blood pressure in 185 whites consuming an isocaloric constant diet with a randomized order of 7 days of low sodium (Na+) and 7 days of high Na+ intake. Salt sensitivity was defined as a ≥7-mm Hg increase in mean arterial pressure during a randomized transition between low and high Na+ diet.

A total of 35 polymorphisms in 17 candidate genes were assayed, 25 of which were tested for association. Association analyses with salt sensitivity revealed 3 variants that associated with salt sensitivity. Of these, 2 SNPs in SLC4A5 (rs7571842 and rs10177833) demonstrated highly significant results and large effects sizes, using logistic regression. These 2 SNPs had P values of 1.0×10-4 and 3.1×10-4 with odds ratios of 0.221 and 0.221 in unadjusted regression models, respectively, with the G allele at both sites conferring protection. These SNPs remained significant after adjusting for body mass index and age (P=8.9×10-5 and 2.6×10-4 and odds ratios 0.210 and 0.286, respectively). Furthermore, the association of these SNPs with salt sensitivity was replicated in a second hypertensive population. Meta-analysis demonstrated significant associations of both SNPs with salt sensitivity (rs7571842 [P=1.2×10-5]; rs1017783 [P=1.1×10-4]).

In conclusion, SLC4A5 variants are strongly associated with salt sensitivity of blood pressure in 2 separate white populations.

DETAILED DESCRIPTION:
Subjects are placed on an isocaloric diet, one week with high sodium(300mEq) and one week with low sodium(10mEq), in randomized order. Twenty-four hour urine sodium and urine creatinine levels verify diet compliance. Blood pressure measurements are recorded during each diet week by automated blood pressure monitoring system. Each blood pressure is taken in the right arm 3 times while the subject is sitting quietly for 45 minutes .

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-70 (inclusive)
* Sex Male and female
* Race Caucasian and African-American/black
* BMI 18.-0-29.9
* BP Normal

Exclusion Criteria:

* hypertension
* blood pressure > 140/90 mmHg

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2005-01; Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Blood pressure; Change in Mean Arterial Pressure from low salt diet to high salt diet | Study subjects will be observed 5 times during the 2 week intervention
  The mean arterial pressure that will determine salt sensitivity will be assessed during the last day of the diet week. The study will be stopped for any individual during any visit if there is an average blood pressure of >180/114 mmHg.

SECONDARY OUTCOMES:
Urine sodium | Urine chemistry analysis will be assessed from a 24-hour urine collection on the last day of each diet week.
Genetic analysis for specified genes associated with hypertension | During the screening visit

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Carey, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] http://hyper.ahajournals.org/content/early/2012/09/17/HYPERTENSIONAHA.112.196071.full.pdf